CLINICAL TRIAL: NCT05003947
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Inflammatory Bowel Disease
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for IBD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-8-ATG-11-04
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; Inflammatory Bowel Diseases; stem cell treatment
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of inflammatory bowel disease

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of inflammatory bowel disease (IBD). Patients with IBD will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease requiring chemotherapeutic drugs such as methotrexate, an autologous T Cell vaccine will be utilized created from the patient's own T cells obtained by apheresis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease or Ulcerative Colitis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Four year follow-up
  The SIBDQ is a questionnaire to assess the physical, social, emotional, and systemic status for IBD patients. It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

REFERENCES:
- [Background] Jowett SL, Seal CJ, Barton JR, Welfare MR. The short inflammatory bowel disease questionnaire is reliable and responsive to clinically important change in ulcerative colitis. Am J Gastroenterol. 2001 Oct;96(10):2921-8. doi: 10.1111/j.1572-0241.2001.04682.x. PMID 11693327
- [Background] Wilcox AR, Dragnev MC, Darcey CJ, Siegel CA. A new tool to measure the burden of Crohn's disease and its treatment: do patient and physician perceptions match? Inflamm Bowel Dis. 2010 Apr;16(4):645-50. doi: 10.1002/ibd.21094. PMID 19714751
- [Background] Hu J, Zhao G, Zhang L, Qiao C, Di A, Gao H, Xu H. Safety and therapeutic effect of mesenchymal stem cell infusion on moderate to severe ulcerative colitis. Exp Ther Med. 2016 Nov;12(5):2983-2989. doi: 10.3892/etm.2016.3724. Epub 2016 Sep 20. PMID 27882104
- [Background] Zhang J, Lv S, Liu X, Song B, Shi L. Umbilical Cord Mesenchymal Stem Cell Treatment for Crohn's Disease: A Randomized Controlled Clinical Trial. Gut Liver. 2018 Jan 15;12(1):73-78. doi: 10.5009/gnl17035. PMID 28873511